CLINICAL TRIAL: NCT02694575
Title: The Impact of Glucose Lowering Therapies Including Dipeptidyl Peptidase-4 Inhibitor on Circulating Endothelial Progenitor Cells (EPCs) and Its Mobilising Factor Stromal Derived Factor-1α (SDF-1α) in Patients With Type 2 Diabetes
Brief Title: The Impact of Glucose Lowering Therapies on Circulating Endothelial Progenitor Cells and Its Mobilising Factor Stromal Derived Factor-1α in Patients With Type 2 Diabetes
Acronym: IGLOOS
Status: Completed | Type: Observational
Sponsor: University of Leicester (Other)
Collaborators: University Hospitals, Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 0483
Record Dates: First submitted 2016-02-23; First posted 2016-02-29 (Estimated); Last update posted 2020-01-30 (Actual); Status verified 2018-05

CONDITIONS: Diabetes Mellitus, Type 2; Cardiovascular Diseases
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Peripheral Blood Mononuclear Cells (PBMCs) for subsequent EPC quantification:
  PBMCs will be isolated from venous blood collected into a 9.7ml sodium heparin blood tube. EPCs will be quantified as cells showing dual positivity for the cell surface / transmembrane markers: CD24 and KDR (Kinase Insert Domain Receptor). SDF-1α analysis and the analysis of biomarkers associated with the prevalence of circulating EPCs will be measured using sandwich ELISA and multi-array ELISA technology in-line with manufacturer protocols. Analysis of endogenous DPP4 will be assayed using a commercial colorimetric assay; again manufacturer protocols will be followed. Biomarker and DPP4 analysis will be carried out in one batch on stored sodium heparin plasma samples.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Other: Other - currently on other treatment (i.e., non-incretin based therapies)
- GLP-1: Currently on GLP-1 analogue therapy
- DPP-4: Currently on DPP-4 inhibitor therapy

SUMMARY:
This is a cross-sectional observational study aiming to examine and compare the impact of incretin based therapies i.e. dipeptidyl peptidase-4 (DPP4) inhibitors and glucagon-like peptide-1 (GLP-1) analogues, on endothelial progenitor cells (EPCs) and its mobilising factor, stromal derived factor-1 α (SDF-1 α), in patients with type 2 diabetes mellitus (T2DM) who are well established on those treatments. EPCs provide vascular protection by means of endothelial repair and neogenesis. This endothelial protective effect may potentially benefit patients affected by micro or macrovascular complications arising from vascular injury e.g. cardiovascular disease in T2DM. The study is of particular interest as a small study has shown an increase in level of circulating EPC in patients treated with DPP-4 inhibitors, thought to be mediated via the up regulation of its mobilising factor SDF-1 α.

DETAILED DESCRIPTION:
Diabetes is a chronic condition reported to affect 366 million people globally in 2011 and estimated to rise to 552 million by 2030 worldwide, i.e. one in 10 adults. In the UK alone, the prevalence is 4.5% and approximately 5 million people are projected to be affected in 2025. Of the entire population of people with diabetes, Type 2 Diabetes Mellitus (T2DM) constitutes more than 90%. In the United Kingdom Prospective Diabetes Study (UKPDS), 50% of the people with T2DM presented with micro and/or macrovascular complications at the time of diagnosis. It is well established that people with T2DM also have 4 to 5 times greater risk of cardiovascular complications compared to the general population, accounting for 80% of mortality. Thus, the burden of diabetes and its associated complications on health care services are enormous. Prescribing medications for the complications associated with diabetes alone costs 3 to 4 times more than the cost of medications for managing diabetes in the National Health Service (NHS). Thus, therapies that simultaneously target glycaemic control and diabetic complications particularly cardiovascular disease (CVD) independent of their glucose lowering effect are desirable.

The current study aims to evaluate the therapeutic effects of incretin based therapies (DPP-4 inhibitors versus GLP-1 analogues) and incretin based therapies versus non-incretin based treatments on levels of EPCs, SDF-1α and other biomarkers in patients with T2DM established on these treatments (receiving for >3 months).

Study objectives To investigate if treatment with DPP-4 inhibitors in patients with T2DM is associated with increased levels of Endothelial Progenitor Cells (EPCs) and Stromal Derived Factor-1 α (SDF-1α) compared to those receiving GLP-1 analogues in a cross sectional analysis adjusted for confounders.

Further, the study aims to determine if treatment with incretin based therapies is associated with higher circulating levels of EPC and SDF1-α compared to non-incretin based therapies.

Preparation of Peripheral Blood Mononuclear Cells (PBMCs) for subsequent EPC quantification PBMCs will be collected using standard techniques. In brief PBMCs will be isolated from venous blood collected into a 9.7ml sodium heparin blood tube (which will subsequently be stored at room temperature for up to 4 hours). The blood samples will then be centrifuged (1500g for 10 min at 4⁰C) and the plasma layer will be collected for later biomarker analysis (aliquots of plasma will be frozen at -80⁰C until use). The buffy coat layer (the white opaque layer that lies directly above the red cell pellet) will be used for PBMC isolation. To isolate the PBMCs, the buffy coat will be centrifuged at 400g on a Ficoll gradient (1.077g/ml) for 30 minutes and the resulting cellular layer will then undergo 3 further washes (300g for 10 minutes and 20g for 10 minutes X2) to wash the cells and deplete platelets. To calculate the number of PBMC isolated, the pellet will be suspended in a known volume of Phosphate Buffered Solution (PBS) (1ml) and a small quantity (10µl) will be assessed for quantity and viability under an inverted microscope using a haemocytometer and a vital stain (Trypan blue).

To prevent inter-assay variation due to longitudinal sample collection, the samples will be stored in liquid nitrogen vapour (using standard freezing protocols) and quantification of the EPCs will be performed as one batch on the stored samples.

Quantification of EPC EPCs will be quantified as cells showing dual positivity for the cell surface / transmembrane markers: Cluster of Differentiation 24 (CD24) and Kinase Domain Receptor (KDR). Standardized flow cytometry protocols will be employed. In brief, the cells will be thawed and immunofluorescent cell staining will be performed using the fluorescent conjugated antibodies: CD34-fluorescein isothiocyanate (FITC) and KDR-phycoerythrin (PE). For each patient, a corresponding negative control with IgG2a-FITC-PE will be processed. The number of circulating EPCs will be expressed in terms of the total number of cells displaying dual positivity for CD24 and KDR per µl blood originally processed.

Biomarkers SDF-1α analysis and the analysis of biomarkers associated with the prevalence of circulating EPCs will be measured using sandwich ELISA and multi-array ELISA technology in-line with manufacturer protocols. Analysis of endogenous DPP4 will be assayed using a commercial colorimetric assay; again manufacturer protocols will be followed. Biomarker and DPP4 analysis will be carried out in one batch on stored sodium heparin plasma samples.

Statistics Statistical methods and analysis Baseline characteristics will be displayed by group (those currently receiving DPP-4 inhibitor, those currently receiving GLP-1analogue, and those currently not using DPP-4 inhibitor or GLP-1 analogue) as mean and standard deviation for normally distributed continuous variables, median and interquartile range for non-normally distributed continuous variables, and counts and percentages for categorical variables. The primary outcome (EPC) will be compared by treatment group using linear regression, with and without adjustment for potential confounders. The confounders to be considered are age, gender, ethnicity, body mass index, duration of T2DM and insulin treatment. The mean EPC and its 95% confidence interval in each of the three groups will be presented as well as the mean difference between DPP-IV vs GLP-1 treatment group and between incretin vs non-incretin treatment groups. A similar analysis will be used for all continuous secondary outcomes. Binary outcomes will be compared by groups using logistic regression analysis with and without adjustment for the same confounders. All statistical tests will be 2 sided and p<0.05 will be taken to be statistically significant.

Sample size Based on the power of 80% and significance at 0.025 (to allow for two primary comparisons, i.e. DPP-IV vs GLP-1 users and incretin users vs non-incretin users), 216 patients (72 in each of the three groups) will be required to detect a difference of 10 EPC/μl assuming a SD of 19.2 to the power of 24. This sample size will also allow a difference of 8 pg/ml of SDF-1α to be detected with 75% power assuming a SD of 16 to the power of 24.

Data management Data collection sheet management All clinical data will be stored in a secure area at the Leicester Diabetes Centre. Each enrolled subject will be allocated a unique study identification number (ID) so that the electronic database remains anonymous.

The Data Collection Form (Case report Form, CRF) is the primary data collection instrument. Data management check will take place and missing data will be explained where possible. If the item is not applicable to the individual case, N/A will be written. All entries will be printed legibly in black ink. If any entry error has been made, to correct the error, a single line will be drawn through the incorrect entry and the correct data entered above it. All such changes will be initialled and dated. For clarification of illegible or uncertain entries, the clarification will be printed above the item and this will be initialled and dated.

Documentation storage, access, security, archiving All study documentation containing identifiable patient data will be managed in accordance with International Conference on Harmonisation-Good Clinical Practice (ICH-GCP), Research Governance Framework for Health and Social Care and the Data Protection Act. Information will only be obtained from the patient if necessary for the study.

All electronic data will be stored on secure university (University of Leicester) or hospital (University Hospitals of Leicester NHS Trust) network drives, to which only the relevant study staff have access, which is granted by the research team.

All study documents and data will be kept for 5 years or the minimum determined by the regulatory authorities, whichever is longer. The study file will be archived in line with the Trust policy.

Data confidentiality Each participant will be assigned a unique identification number upon recruitment. Patients' contact details will be held on a separate database and used to arrange study visits. The database will be password protected and only members of the research team contacting patients will have access. All data collected during the study will be stored anonymously on a separate database. Again access will be password protected and restricted to relevant members of the research team. Electronic data will be stored in the University or NHS system.

Safety Issues The Investigators do not foresee any adverse events over and above those associated with everyday life and routine health care that could be attributable to the study. The study involves only one venepuncture to withdraw venous blood and hence carries a very low risk of having untoward effects. However, all participants will undergo venepuncture which can occasionally result in bruising, swelling and temporary discomfort.

The Investigators will follow the University of Leicester guidelines for managing and reporting a Serious Adverse Event (SAE) or Suspected Unexpected Serious Adverse Reaction (SUSAR), which follow those outlined in Good Clinical Practice (GCP) guidance.

A SAE is any adverse event or unexpected adverse reaction that results in death is life-threatening requires hospitalisation or prolongation of existing hospitalisation results in persistent or significant disability or incapacity consists of a congenital anomaly or birth defect. In addition, the Investigators will also define an event as serious if it is an important and significant medical event that may not be immediately life threatening or resulting in death or hospitalisation but, based upon appropriate medical judgement may jeopardise the patient or may require intervention to prevent one or more outcomes listed above. Adverse events which do not fall into these categories are defined as non-serious.

All SAEs will be reported internally to the University Hospitals of Leicester (UHL) NHS Trust Research & Development (R&D) and the sponsor (University of Leicester) using appropriate reporting forms, within 24 hours of the study team becoming aware of the event. The principal investigator is responsible for the review and submission of any SAE, or in their absence, another member of the team (in order to avoid a delay). The investigator site file will contain documentation for SAE reports and evidence of timely submissions.

ELIGIBILITY:
Inclusion Criteria:

* Capacity to provide informed consent before any study-related activities
* Individuals aged 35-70 years inclusive
* Both male and female
* Diagnosed with T2DM for at least 1 year
* On DPP4-inhibitor, GLP-1 analogue or non-incretin agent for at least 3 months regardless of their background treatment
* White European or South Asian ethnicity (to increase the comparability of treatment groups)

Exclusion Criteria:

* Type 1 diabetes
* Individuals <35 or >70 years of age
* Prescribed thiazolidinediones or sodium-glucose co-transporter-2 (SGLT-2) inhibitors within the last 3 months
* Any form of terminal illness

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients aged between 35 and 70 years of age (inclusve) who have established Type 2 Diabetes mellitus (T2DM) and who have been receiving either (a) DPP-4 inhibitors, (b) GLP-1 analogues, or (c) non-incretin based treatments for at least 3 months (or more).
Sampling Method: Non-Probability Sample
Enrollment: 241 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2017-04-12 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
EPC | Single sample analysis - no time frame
  The measure of number of circulating Endothelial Progenitor Cells (EPCs) (EPC/μl)

SECONDARY OUTCOMES:
SDF 1-α (Stromal derived factor-1α) | Single sample analysis - no time frame
  Level of SDF 1-α (Stromal derived factor-1α) biomarker analysis
Glucagon-like peptide 1 (GLP-1) | Single sample analysis - no time frame
  Level of GLP 1 (Glucagon like peptide 1) biomarker analysis.
Dipeptidyl peptidase 4 (DDP-4) | Single sample analysis - no time frame
  Level of DPP 4 (Dipeptidyl peptidase 4) biomarker analysis.
C-reactive protein | Single sample analysis - no time frame
  Level of C-reactive protein biomarker analysis.
Nitric oxide (NO) | Single sample analysis - no time frame
  Level of NO (Nitric oxide) biomarker analysis.
Hypoxia-inducible factor -1α (HIF-1α) | Single sample analysis - no time frame
  Level of HIF -1α (Hypoxia inducible factor -1α) biomarker analysis.
Vascular endothelial growth factor (VEGF) | Single sample analysis - no time frame
  Level of VEGF (Vascular endothelial growth factor) biomarker analysis.
Granulocyte colony stimulating factor (G-CSF) | Single sample analysis - no time frame
  Level of G-CSF (Granulocyte colony stimulating factor) biomarker analysis.
Stem cell factor (SCF) | Single sample analysis - no time frame
  Level of SCF (Stem cell factor) biomarker analysis.
High Mobility Group Box-1 (HMGB-1) | Single sample analysis - no time frame
  Level of HMGB-1 (high mobility group box-1) biomarker analysis.
Full blood count | Single sample analysis - no time frame
  Full blood count analysis
HbA1c | Single sample analysis - no time frame
  HbA1c analysis
Renal function | Single sample analysis - no time frame
  Renal function analysis

CONTACTS AND LOCATIONS:
Overall Officials: Melanie J Davies, MBBS MD, Principal Investigator — University of Leicester
Locations (1):
- Leicester Diabetes Centre, Leicester, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Clinically significant blood result data will be shared with the participant's General Practitioner when appropriate.

REFERENCES:
- [Background] IDF. IDF diabetes atlas 5th Edition. 2011.
- [Background] DUK. Diabetes in the UK 2010 Key Satistics on Daibetes. 2010: 1-21.
- [Background] Turner RC, Holman RR. Lessons from UK prospective diabetes study. Diabetes Res Clin Pract. 1995 Aug;28 Suppl:S151-7. doi: 10.1016/0168-8227(95)01105-m. PMID 8529508
- [Background] Buse JB, Ginsberg HN, Bakris GL, Clark NG, Costa F, Eckel R, Fonseca V, Gerstein HC, Grundy S, Nesto RW, Pignone MP, Plutzky J, Porte D, Redberg R, Stitzel KF, Stone NJ; American Heart Association; American Diabetes Association. Primary prevention of cardiovascular diseases in people with diabetes mellitus: a scientific statement from the American Heart Association and the American Diabetes Association. Diabetes Care. 2007 Jan;30(1):162-72. doi: 10.2337/dc07-9917. PMID 17192355
- [Background] Nauck M, Stockmann F, Ebert R, Creutzfeldt W. Reduced incretin effect in type 2 (non-insulin-dependent) diabetes. Diabetologia. 1986 Jan;29(1):46-52. doi: 10.1007/BF02427280. PMID 3514343
- [Background] Nauck MA, Vardarli I, Deacon CF, Holst JJ, Meier JJ. Secretion of glucagon-like peptide-1 (GLP-1) in type 2 diabetes: what is up, what is down? Diabetologia. 2011 Jan;54(1):10-8. doi: 10.1007/s00125-010-1896-4. Epub 2010 Sep 25. PMID 20871975
- [Background] Drucker DJ, Nauck MA. The incretin system: glucagon-like peptide-1 receptor agonists and dipeptidyl peptidase-4 inhibitors in type 2 diabetes. Lancet. 2006 Nov 11;368(9548):1696-705. doi: 10.1016/S0140-6736(06)69705-5. PMID 17098089
- [Background] Derosa G, Maffioli P, Salvadeo SA, Ferrari I, Ragonesi PD, Querci F, Franzetti IG, Gadaleta G, Ciccarelli L, Piccinni MN, D'Angelo A, Cicero AF. Exenatide versus glibenclamide in patients with diabetes. Diabetes Technol Ther. 2010 Mar;12(3):233-40. doi: 10.1089/dia.2009.0141. PMID 20151774
- [Background] Arakawa M, Mita T, Azuma K, Ebato C, Goto H, Nomiyama T, Fujitani Y, Hirose T, Kawamori R, Watada H. Inhibition of monocyte adhesion to endothelial cells and attenuation of atherosclerotic lesion by a glucagon-like peptide-1 receptor agonist, exendin-4. Diabetes. 2010 Apr;59(4):1030-7. doi: 10.2337/db09-1694. Epub 2010 Jan 12. PMID 20068138
- [Background] Nikolaidis LA, Mankad S, Sokos GG, Miske G, Shah A, Elahi D, Shannon RP. Effects of glucagon-like peptide-1 in patients with acute myocardial infarction and left ventricular dysfunction after successful reperfusion. Circulation. 2004 Mar 2;109(8):962-5. doi: 10.1161/01.CIR.0000120505.91348.58. Epub 2004 Feb 23. PMID 14981009
- [Background] Sokos GG, Nikolaidis LA, Mankad S, Elahi D, Shannon RP. Glucagon-like peptide-1 infusion improves left ventricular ejection fraction and functional status in patients with chronic heart failure. J Card Fail. 2006 Dec;12(9):694-9. doi: 10.1016/j.cardfail.2006.08.211. PMID 17174230
- [Background] Thrainsdottir I, Malmberg K, Olsson A, Gutniak M, Ryden L. Initial experience with GLP-1 treatment on metabolic control and myocardial function in patients with type 2 diabetes mellitus and heart failure. Diab Vasc Dis Res. 2004 May;1(1):40-3. doi: 10.3132/dvdr.2004.005. PMID 16305055
- [Background] Asahara T, Murohara T, Sullivan A, Silver M, van der Zee R, Li T, Witzenbichler B, Schatteman G, Isner JM. Isolation of putative progenitor endothelial cells for angiogenesis. Science. 1997 Feb 14;275(5302):964-7. doi: 10.1126/science.275.5302.964. PMID 9020076
- [Background] Werner N, Kosiol S, Schiegl T, Ahlers P, Walenta K, Link A, Bohm M, Nickenig G. Circulating endothelial progenitor cells and cardiovascular outcomes. N Engl J Med. 2005 Sep 8;353(10):999-1007. doi: 10.1056/NEJMoa043814. PMID 16148285
- [Background] Jialal I, Fadini GP, Pollock K, Devaraj S. Circulating levels of endothelial progenitor cell mobilizing factors in the metabolic syndrome. Am J Cardiol. 2010 Dec 1;106(11):1606-8. doi: 10.1016/j.amjcard.2010.07.039. Epub 2010 Sep 21. PMID 21040691
- [Background] Fadini GP, Miorin M, Facco M, Bonamico S, Baesso I, Grego F, Menegolo M, de Kreutzenberg SV, Tiengo A, Agostini C, Avogaro A. Circulating endothelial progenitor cells are reduced in peripheral vascular complications of type 2 diabetes mellitus. J Am Coll Cardiol. 2005 May 3;45(9):1449-57. doi: 10.1016/j.jacc.2004.11.067. PMID 15862417
- [Background] Tepper OM, Galiano RD, Capla JM, Kalka C, Gagne PJ, Jacobowitz GR, Levine JP, Gurtner GC. Human endothelial progenitor cells from type II diabetics exhibit impaired proliferation, adhesion, and incorporation into vascular structures. Circulation. 2002 Nov 26;106(22):2781-6. doi: 10.1161/01.cir.0000039526.42991.93. PMID 12451003
- [Background] Hill JM, Zalos G, Halcox JP, Schenke WH, Waclawiw MA, Quyyumi AA, Finkel T. Circulating endothelial progenitor cells, vascular function, and cardiovascular risk. N Engl J Med. 2003 Feb 13;348(7):593-600. doi: 10.1056/NEJMoa022287. PMID 12584367
- [Background] Vasa M, Fichtlscherer S, Aicher A, Adler K, Urbich C, Martin H, Zeiher AM, Dimmeler S. Number and migratory activity of circulating endothelial progenitor cells inversely correlate with risk factors for coronary artery disease. Circ Res. 2001 Jul 6;89(1):E1-7. doi: 10.1161/hh1301.093953. PMID 11440984
- [Background] Kunz GA, Liang G, Cuculi F, Gregg D, Vata KC, Shaw LK, Goldschmidt-Clermont PJ, Dong C, Taylor DA, Peterson ED. Circulating endothelial progenitor cells predict coronary artery disease severity. Am Heart J. 2006 Jul;152(1):190-5. doi: 10.1016/j.ahj.2006.02.001. PMID 16824855
- [Background] Schmidt-Lucke C, Rossig L, Fichtlscherer S, Vasa M, Britten M, Kamper U, Dimmeler S, Zeiher AM. Reduced number of circulating endothelial progenitor cells predicts future cardiovascular events: proof of concept for the clinical importance of endogenous vascular repair. Circulation. 2005 Jun 7;111(22):2981-7. doi: 10.1161/CIRCULATIONAHA.104.504340. Epub 2005 May 31. PMID 15927972
- [Background] Fadini GP, Sartore S, Agostini C, Avogaro A. Significance of endothelial progenitor cells in subjects with diabetes. Diabetes Care. 2007 May;30(5):1305-13. doi: 10.2337/dc06-2305. Epub 2007 Feb 2. No abstract available. PMID 17277037
- [Background] Ahren B, Landin-Olsson M, Jansson PA, Svensson M, Holmes D, Schweizer A. Inhibition of dipeptidyl peptidase-4 reduces glycemia, sustains insulin levels, and reduces glucagon levels in type 2 diabetes. J Clin Endocrinol Metab. 2004 May;89(5):2078-84. doi: 10.1210/jc.2003-031907. PMID 15126524
- [Background] Fadini GP, Boscaro E, Albiero M, Menegazzo L, Frison V, de Kreutzenberg S, Agostini C, Tiengo A, Avogaro A. The oral dipeptidyl peptidase-4 inhibitor sitagliptin increases circulating endothelial progenitor cells in patients with type 2 diabetes: possible role of stromal-derived factor-1alpha. Diabetes Care. 2010 Jul;33(7):1607-9. doi: 10.2337/dc10-0187. Epub 2010 Mar 31. PMID 20357375